CLINICAL TRIAL: NCT06136390
Title: OXYMIND: Oxytocin-augmented Group Psychotherapy for Patients With Schizophrenia
Acronym: OXYMIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Kerem Böge, PD Dr. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 401743
Record Dates: First submitted 2023-11-04; First posted 2023-11-18 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia Spectrum Disorders
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Active Comparator): The patients received a spray of the synthetic oxytocin (24 I.U. Syntocinon®) in combination with mindfulness-based group therapy (MBGT) over 4 weeks once a week. Due to an effect latency of 30-80 mins after intranasal administration of oxytocin on social behavior, the dose was administered 45 min before the 50-min session.
  Interventions: Other: Oxytocin
- Placebo (Placebo Comparator): The patients received a spray of placebo (24 I.U. Syntocinon®) in combination with mindfulness-based group therapy (MBGT) over 4 weeks once a week. Due to an effect latency of 30-80 mins after intranasal administration of oxytocin on social behavior, the dose was administered 45 min before the 50-min session.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Oxytocin — Oxytocin nasal spray in combination with mindfulness based group therapy (MBGT).
  Arms: Oxytocin
Other: Placebo — Placebo nasal spray in combination with mindfulness based group therapy (MBGT).
  Arms: Placebo

SUMMARY:
The effectiveness of current treatment options for sociocognitive deficits and negative symptoms (NS) in schizophrenia spectrum disorders (SSD) remains limited. The cause of NS is thought to be an interference between the mesocorticolimbic dopamine system for social reward expectancy and the network for socioemotional processes. Oxytocin (OXT) may enhance functional connectivity between these neuronal networks. Lower plasma OXT levels correlate negatively with NS severity and deficits in social cognition in SSD. It has been shown that intranasal OXT administration improves social cognition in healthy subjects but in SSD results are inconsistent. According to the social salience hypothesis, the effect of OXT varies depending on the social context and individual factors. Also, OXT-mediated effects on psychopathology and NS may depend on genetic variants of OXT receptors (OXTR). In a pilot study, the investigators demonstrated a lower NS by OXT administration in the positive social context of MBGT in SSD. The investigators also demonstrated that NS and other symptoms improved after mindfulness-based group psychotherapy (MBGT). The aim of this study in individuals with SSD is to examine the effect of combining OXT administration with MBGT on NS, affect, and stress with psychological and biological markers. The main hypothesis to be tested is that the use of OXT compared to placebo prior to MBGT in patients with SSD will result in a greater reduction in NS. The research design is based on an experimental, triple-blind, randomized, placebo-controlled trial.

DETAILED DESCRIPTION:
Schizophrenia spectrum disorders (SCZ) are severe mental illnesses with a lifetime prevalence of 1-2%. Three core syndromes characterize SCZ: positive and negative syndromes (NS), as well as a cognitive syndrome. The effectiveness of current treatment options for negative symptoms (NS) and sociocognitive deficits in schizophrenia spectrum disorders (SSD) remains limited.

The cause of NS is thought to be an interference between the mesocorticolimbic dopamine system for social reward expectancy and the network for socioemotional processes. Oxytocin (OXT) may enhance functional connectivity between these neuronal networks. Lower plasma OXT levels correlate negatively with NS severity and deficits in social cognition in SSD. It has been shown that intranasal OXT administration improves social cognition in healthy subjects but in SSD results are inconsistent. According to the social salience hypothesis, the effect of OXT varies depending on the social context and individual factors. Also, OXT-mediated effects on psychopathology and NS may depend on genetic variants of OXT receptors (OXTR). In a pilot study, the investigators demonstrated lower NS by OXT administration in a positive social context of MBGT in SSD. The investigators also demonstrated that NS and other symptoms improved after mindfulness-based group psychotherapy (MBGT).

The aim of this study in individuals with SSD is to examine the effect of combining OXT administration with MBGT on NS, affect, and stress. The main hypothesis to be tested is that the use of OXT compared to placebo prior to MBGT in patients with SSD will result in a greater reduction in NS, i.e. the difference in T7 - T0 of the negative syndrome subscale of the PANSS (Positive and Negative Syndrome Scale) after 4 weeks. The PANSS as a validated and structured clinical interview will be collected by a blinded psychiatrist. MBGT - sessions by experienced psychotherapists take place over four weeks. These sessions as a positive social context take place once a week in a group of about six patients. Participants received either synthetic oxytocin or a placebo 30 minutes before MBGT.

The role of genetic variations (OXTR genes) for the treatment effect on NS will be explored too as well as the effect on various stress markers including cortisol levels and the endocannabinoid system, affect, group cohesion and mindfulness.

The research design is based on an experimental, triple-blind, randomized, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* declaration of consent
* Psychiatric diagnosis of schizophrenia (ICD-10: F2x.x spectrum) for group of patients
* Mild to moderate positive symptoms (5 ≤ Positive symptoms on individual items using P- PANSS)
* German should either be the native language or spoken at a native level.
* No change in systematically recorded psychopharmacological medication in the last 2 weeks before study inclusion.

Exclusion Criteria:

* Acute psychotic episode with severe positive symptoms (ICD-10: F2 spectrum, 6 ≥ positive symptoms on individual items using P-PANSS).
* Acute suicidality
* Acute consumption phase of a substance dependence, except nicotine
* No severe physical impairments, neurological diseases and e.g. severe craniocerebral trauma e.g. early childhood brain damage
* Pregnancy and breastfeeding
* Current electroconvulsive therapy

If one of the following criteria applies to the participants, we will conduct an individual consultation in advance to determine whether participation in the study is possible:

* Overweight or underweight (body mass index (BMI) < 17.5 or > 30)
* Disease of the endocrine system
* Impaired kidney or liver function
* Metabolic diseases
* Asthma
* Change in blood potassium or sodium levels

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Change in PANSS Negative Symptoms | Baseline (T0), post-intervention at week 4 (T4) and follow-up (week 8, T5)
  The Positive and Negative Syndrome Scale (PANSS) is one of the most widely used rater instruments for the assessment of the presence and severity of psychotic symptoms. Each scale comprises seven statements which are rated by the interviewer using a seven-point Likert format (from 1= absent to 7= extreme). The PANSS is reported to have satisfactory internal consistency, good interrater reliability and construct validity.

SECONDARY OUTCOMES:
Change and group differences in BNSS Brief Negative Symptom Scale | Baseline (T0), post-intervention at week 4 (T7) and follow-up (week 8, T8)
  The Brief Negative Symptom Scale (BNSS) is a 13-item rater-based instrument designed for clinical trials and other studies that measures 5 domains: blunted affect, alogia, asociality, anhedonia, and avolition. The interrater, test-retest, and internal consistency of the instrument were strong, with respective intraclass correlation coefficients of 0.93 for the BNSS total score and values of 0.89-0.95 for individual subscales.
Change and group differences in SNS Negative Symptoms | Baseline (T0), post-intervention at week 2 (T3), post-intervention at week 4 (T9) and follow-up (week 8, T5)
  This is a 20-item self-reported questionnaire with five subscales, namely alogia, avolition, anhedonia, social withdrawal and diminished emotional range. These subscales cluster on two factors, the apathy and emotional components. Participants can estimate the answer to each question on a scale from 0 (strongly disagree) to 3 (strongly agree). The scale was shown to have good internal consistency with Cronbach's alpha = .87.
Change and group differences in CDSS Calgary Depression Scale of Schizophrenia | Baseline (T0), post-intervention at week 4 (T7) and follow-up (week 8, T8)
  The Calgary Depression Scale for Schizophrenia (CDSS) is a nine item clinician rated outcome measure that assesses the level of depression in people with schizophrenia. It is the only depression scale designed to assess depression in people with a schizophrenia spectrum disorder. It distinguishes depressive symptoms from negative symptoms and is sensitive to change.
Change and group differences in cortisol saliva levels | Baseline (T0), pre- and post-intervention in week 1 - 4 (T1-T7) and follow-up (week 8, T5)
  Saliva samples will be taken before and after each MBGT session to determine Cortisol saliva levels
Change and group differences in DASS-21 Depression, Anxiety, and Stress Scale | aseline (T0), post-intervention at week 2 (T3), post-intervention at week 4 (T7) and follow-up (week 8, T9)
  The 21-item Depression, Anxiety, and Stress Scale (DASS-21) is assessed on a four-point Likert-scale ranging from (0) "did not apply to me at all over the last week" to (3) "applied to me very much last week." It shows internal consistencies of α > 0.80 across the three subscales and has shown to be a useful measurement tool for patients with SSD.
Change and group differences in stress via visual analogue scale (Bubbles) | Baseline (T0), pre- and post-intervention in week 1 - 4 (T1-T7) and follow-up (week 8, T8)
  Stress via visual analogue scale. Self-rating instrument to measure stress through four items on a seven-point Likert-scale ranging from "not at all" (0) to "extreme" (6) visualized through bubbles increasing in size.
Change and group differences in PANAS (Positive and Negative Affect Scale) | Baseline (T0), pre- and post-intervention in week 1 - 4 (T1-T7) and follow-up (week 8, T8)
  The PANAS contains 20 items, each consisting of an adjective describing an emotion. The participants have to select how applicable this adjective is to their current state from 1 (not at all) to 5 (extremely). Ten items are assigned to the positive (e.g. "Excited") as well as the negative scale (e.g. "Fearful"). The reliability of the PANAS ranges from .86 to .93.
Change and group differences in PSP Social Functioning | Baseline (T0), post-intervention at week 4 (T7) and follow-up (week 8, T8)
  The Personal and Social Performance Scale (PSP) is a rater-based questionnaire used to assess social functioning in patients with SSD. The PSP showed good test-retest reliability (ICC = 0.79) in patients with schizophrenia.
Change and group differences in SMQ Mindfulness | Baseline (T0), post-intervention at week 4 (T7) and follow-up (week 8, T8)
  The SMQ comprises 16 items that are rated on a seven-point Likert-scale ranging from (6) "agree totally" to (0) "disagree totally". Consequently, the total score ranges from 0 to 96, with a higher score indicating higher mindfulness. The internal consistency of the German version of the SMQ was Cronbach's α = 0.89.
Change and group differences in GCQ-S Group Climate Questionnaire (Short Version) | Post-intervention at week 1-4 (T1-T7)
  The GCQ-S is a 12 item questionnaire designed to assess individual group members' perceptions of the group's therapeutic environment. It consists of three domains: Engaged, conflict and avoiding and will be used as a self-report, such as a rater-based instrument.
Change and group differences in endocannibinoid levels | Baseline (T0), post-intervention week 1 (T1), post-intervention week 4 (T7) and follow-up (week 8, T8)
  Venous blood samples will be taken to determine the endocannibinoid levesls to obtain an individual baseline and comparison level.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Zierhut, MD, Principal Investigator — Charite University, Berlin, Germany; Kerem Böge, PD, Principal Investigator — Charite University, Berlin, Germany; Eric Hahn, PD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boge K, Hahne I, Bergmann N, Wingenfeld K, Zierhut M, Thomas N, Ta TMT, Bajbouj M, Hahn E. Mindfulness-based group therapy for in-patients with schizophrenia spectrum disorders - Feasibility, acceptability, and preliminary outcomes of a rater-blinded randomized controlled trial. Schizophr Res. 2021 Feb;228:134-144. doi: 10.1016/j.schres.2020.12.008. Epub 2021 Jan 9. PMID 33434727